CLINICAL TRIAL: NCT05767398
Title: A Single-dose, Open-label, Randomized, Replicate Crossover Study in Healthy Adult Subjects to Assess the Bioequivalence of a Zanubrutinib Tablet Compared to Zanubrutinib Capsules
Brief Title: Bioequivalence of a Zanubrutinib Tablet Compared to Capsules in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BGB-3111-114
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Zanubrutinib will be administered as a single dose of treatment (tablet) or reference (capsule) on separate occasions.
  Interventions: Drug: Zanubrutinib
- Sequence 2 (Experimental): Zanubrutinib will be administered as a single dose of treatment (tablet) or reference (capsule) on separate occasions.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Administered as a tablet or capsule
  Other Names: BGB-3111; Brukinsa

SUMMARY:
Study to determine the bioequivalence of a zanubrutinib tablet compared to capsules in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m^2, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead ECGs, vital sign measurements, and clinical laboratory evaluations as assessed by the investigator or designee
* Female participants must be of non-childbearing potential (surgically sterile or postmenopausal)

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee
* Evidence of any infections (bacterial, viral, fungal, parasitic, COVID-19) within 4 weeks prior to the first dose of study drug, as determined by the investigator or designee
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator or designee
* History or presence of an abnormal ECG prior to the first dose of the study drug that, in the opinion of the investigator or designee, is clinically significant
* Abnormal liver function tests, as defined by aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin >upper limit of normal (ULN) range
* Positive hepatitis panel and/or positive human immunodeficiency virus test

Note: Other protocol defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Predose and up to 48 hours postdose up to Day 10
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t) | Predose and up to 48 hours postdose up to Day 10
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) | Predose and up to 48 hours postdose up to Day 10
Time of the maximum observed plasma concentration (Tmax) | Predose and up to 48 hours postdose up to Day 10
Apparent terminal elimination half-life (t1/2) | Predose and up to 48 hours postdose up to Day 10
Apparent volume of distribution (Vz/F) | Predose and up to 48 hours postdose up to Day 10
Rate of decrease of concentration in the terminal phase (λz) | Predose and up to 48 hours postdose up to Day 10
Apparent oral clearance (CL/F) | Predose and up to 48 hours postdose up to Day 10

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 30 days after last dose; up to approximately 7 weeks
Number of participants with clinically significant laboratory values | Up to 30 days after last dose; up to approximately 7 weeks
  Laboratory values are based on hematology, clinical chemistry, and urinalysis test results
Number of participants with clinically significant electrocardiogram (ECG) results | Up to 30 days after last dose; up to approximately 7 weeks
Number of participants with clinically significant vital sign measurements | Up to 30 days after last dose; up to approximately 7 weeks
  Vital sign measurements include supine blood pressure, supine pulse rate, respiratory rate, and oral body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (1):
- Fortrea Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes